CLINICAL TRIAL: NCT05323227
Title: Association of Lipoprotein (a) With Coronary CTA Assessed High Risk Coronary Disease Attributes and Cardiovascular Outcomes
Brief Title: Lp(a) With CCTA Assessed Parameters and Clinical Outcomes
Acronym: CHART-ACCORD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHART20220404
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with Lp(a) <60mg/dL
  Interventions: Diagnostic Test: Coronary CTA
- Group 2: Patients with Lp(a) ≥60 mg/dL
  Interventions: Diagnostic Test: Coronary CTA

INTERVENTIONS:
Diagnostic Test: Coronary CTA — Patients receive coroanry CTA at the discretion of the physicians in charge. And parameters including plaque burden, minimal lumen area, diameter stenosis, total plaque volume, high-risk plaque characteristics, fractional flow reserve, pullback pressure gradient, fat attenuation index will be analyzed.

SUMMARY:
Lipoprotein(a) [Lp(a)] is a risk factor for cardiovascular events, although the underlying mechanism remains unclear. This study evaluated the relationship between Lp(a) and high-risk attributes (HRA) by coronary computed tomography angiography (CCTA) as well as their prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Lp(a) meaured within 1 week of CCTA examination.

Exclusion Criteria:

* unstable angina pectoris
* acute myocardial infarction
* New York Heart Association class III-IV heart failure
* with a history of bypass surgery
* active infection
* respiratory failure
* chronic kidney disease (estimated glomerular filtration rate [eGFR] <60 ml/min/1.73 m2)
* liver dysfunction (liver enzyme >3 upper reference limit [URL] or bilirubin >2 URL)
* malignancy
* systemic connective tissue disease
* poor CCTA imaging quality not suitable for analysis
* other situations not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable CAD patients with serum Lp(a) measured and underwent CCTA within 1 week at Zhongshan Hospital, Fudan University
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2016-03-20 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Association of Lp(a) level with CCTA measured Parameters | at the index procedure
  Association of Lp(a) level with CCTA measured total plaque volume
Association of Lp(a) level with CCTA measured Parameters | at the index procedure
  Association of Lp(a) level with CCTA measured fractional flow reserve
Association of Lp(a) level with CCTA measured Parameters | at the index procedure
  Association of Lp(a) level with CCTA measured pullback pressure gradient
Association of Lp(a) level with CCTA measured Parameters | at the index procedure
  Association of Lp(a) level with CCTA measured fat attenuation index
Association of Lp(a) level with CCTA measured Parameters | at the index procedure
  Association of Lp(a) level with CCTA measured high-risk plaque characteristics
Major adverse cardiac events | at 24 months from index procedure
  a composite of cardiac death, any myocardial infarction, and stroke

SECONDARY OUTCOMES:
Cardiac death | at 24 months from index procedure
  Cardiac death
Myocardial infarction | at 24 months from index procedure
  Myocardial infarction
Stroke | at 24 months from index procedure
  stroke

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Principal Investigator — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dai N, Hwang D, Lee JM, Zhang J, Jeon KH, Paeng JC, Cheon GJ, Koo BK, Ge J. Feasibility of Quantitative Flow Ratio-Derived Pullback Pressure Gradient Index and Its Impact on Diagnostic Performance. JACC Cardiovasc Interv. 2021 Feb 8;14(3):353-355. doi: 10.1016/j.jcin.2020.10.036. No abstract available. PMID 33541549
- [Background] Shin D, Dai N, Lee SH, Choi KH, Lefieux A, Molony D, Hwang D, Kim HK, Jeon KH, Lee HJ, Jang HJ, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Doh JH, Shin ES, Nam CW, Koo BK, Gwon HC, Ge J, Lee JM. Physiological Distribution and Local Severity of Coronary Artery Disease and Outcomes After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1771-1785. doi: 10.1016/j.jcin.2021.06.013. PMID 34412795
- [Derived] Dai N, Chen Z, Zhou F, Zhou Y, Hu N, Duan S, Wang W, Yu Y, Zhang L, Qian J, Ge J. Association of Lipoprotein (a) With Coronary-Computed Tomography Angiography-Assessed High-Risk Coronary Disease Attributes and Cardiovascular Outcomes. Circ Cardiovasc Imaging. 2022 Dec;15(12):e014611. doi: 10.1161/CIRCIMAGING.122.014611. Epub 2022 Dec 12. PMID 36503252